CLINICAL TRIAL: NCT00256087
Title: The Effect of Prophylactic Probiotic Lactobacilli in Enteral Feeding on Nosocomial Pneumonia Rates in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004.067
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-04

CONDITIONS: Critical Illness
Keywords: Nosocomial rates in critically ill patients
MeSH Terms: conditions — Critical Illness

ARMS (3):
- Standard Care (Placebo Comparator): Two capsules containing placebo will be given 12 hourly
  Interventions: Other: Lactose Powder
- First active treatment (Active Comparator): Two capsules containing probiotic lactobacillus fermentin given 12 hourly
  Interventions: Drug: Probiotic Lactobacillus
- Second active reatment (Active Comparator): Two capsules containing probiotic lactobacillus acidiphilus given 12 hourly
  Interventions: Drug: Probiotic Lactobacillus

INTERVENTIONS:
Drug: Probiotic Lactobacillus
  Arms: First active treatment; Second active reatment
Other: Lactose Powder
  Arms: Standard Care

SUMMARY:
To assess the effect of addition of probiotic Lactobacilli to standard enteral feeding on infection rates and feeding efficacy in critically ill patients.

The study hypothesis is that critically ill patients who receive the addition of probiotic lactobacilli to the enteral feed will lead to a reduced rate of hospital acquired infections.

The null hypothesis is that there will be no significant difference in the rate of hospital acquired infection in critically ill patients who receive enteral feeding with or without the addition of probiotic Lactobacilli.

DETAILED DESCRIPTION:
The patients are randomised to one of three treatment groups. Each comprising of 100 patients.

1. Standard therapy group. Patients will receive enteral feeding (with fibre) aiming at the target feeding rate that is determined by the treating physician and the ICU dietician, as is standard current practice. Two capsule containing placebo will be given 12 hourly via the feeding tube.
2. The first active treatment group, will receive enteral feeding (with fibre) plus probiotic Lactobacillus fermentum included in the feeding regime. Two capsules containing Lactobacillus fermentum (10 11 organisms per capsule) will be delivered via the feeding tube 12 hourly.
3. The second active treatment group will receive enteral feeding (with fibre) plus the probiotic Lactobacillus acidophilus included in the feeding regime. Two capsules containing Lactobacillus acidophilus (2x10 9 organisms per capsule) will be delivered via the feeding tube 12 hourly.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years or over)admitted to ICU with an expected stay of more than 48 hours.
2. Patients who are commenced on enteral feeding via gastric or post pyloric routes.
3. Patients who consent or if the patients is incompetent, their next of kin who consent, to inclusion in the study

Exclusion Criteria:

1. Patients less than 18 years old.
2. Patients who are already receiving probiotic treatment.
3. The lactobacillus acidophilus preparation to be used in the study, contains a very small amount of MSG (total dose of 20mg/day, equivalent to 10% of the initial dose used to test MSG sensitivity) and as a precaution, patients with asthma or recurrent urticaria will be excluded.
4. Patients with HIV infection, pre-existing immunosuppression, or who are pregnant. As the Lactobacillus is a live micro-organism, immunosuppressed and pregnant pateints will be excluded.
5. Patients with a contra-indication to enteral feeding.
6. Patients with contra-indication to placement of enteral feeding tube.
7. Patients or next-of-kin who do not consent to inclusion in the study.
8. Patients who are already enrolled in another study that may influence the outcome of the probiotic study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine if enteral feeding plus probiotic Lactobacilli are associated with a reduced rate of nosocomial pneumonia in critically ill patients. | 28 days

SECONDARY OUTCOMES:
To determine the incidence of complications of enteral feeding with and without added probiotic Lactobacilli. | 28 Days
To assess if the efficacy of enteral feeding in critically ill patients is improved by the addition of probiotic Lactobacilli. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Megan Robertson, Principal Investigator — Intensive Care Unit, Royal Melbourne Hospital
Locations (1):
- Intensive Care Unit Royal Melbourne Hospital Grattan Street, Parkville, Victoria, Australia